CLINICAL TRIAL: NCT01023269
Title: Phase IV, Multi-center, Randomized, Cross-over Study to Demonstrate the Efficacy of Pudendal Neuromodulation for the Treatment of Neurogenic Overactive Bladder
Brief Title: Efficacy Study of Pudendal Neuromodulation for the Treatment of Neurogenic Overactive Bladder
Acronym: ACCEPTANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in the enrolment
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.02.7004
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Neurogenic Overactive Bladder; Urinary Incontinence; Detrusor Overactivity
Keywords: Neurogenic overactive bladder; Urinary incontinence due to incomplete spinal cord injury; Neuromodulation; Neuromodulation for treatment of neurogenic overactive bladder; Patients with Urge urinary incontinence and detrusor overactivity
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ON / OFF (Other): Stimulation ON for 4 weeks, followed by stimulation OFF for 4 weeks.
  Interventions: Device: InterStim Therapy
- OFF / ON (Other): Stimulation OFF for 4 weeks, followed by stimulation ON for 4 weeks.
  Interventions: Device: InterStim Therapy

INTERVENTIONS:
Device: InterStim Therapy — Neuromodulation therapy which delivers low level electrical stimulation to bladder wall for the treatment of overactive bladder with urinary incontinence.

SUMMARY:
The study is designed to demonstrate that treatment with low level stimulation of the bladder muscles reduces symptoms of urinary incontinence in comparison with no stimulation.

DETAILED DESCRIPTION:
The Medtronic InterStim device delivers stimulation therapy for the treatment of chronic intractable (functional) disorders of the pelvis and lower urinary or intestinal tract through the sacral nerve or the pudendal nerve systems.

This trial is designed to demonstrate that neuromodulation of the pudendal nerve will effectively treat patients with neurogenic overactive bladder. Symptoms of urinary incontinence are compared when stimulation is switched on for 4 weeks to stimulation switched off for 4 weeks. After the eight week crossover period, all patients receive treatment and are followed up within the study for 12 months post implant.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete upper motor neuron lesion
* Detrusor overactivity
* Two leaks or two notices of leaks per day
* Mean functional bladder capacity (volume voided per episode) of ≥100 ml

Exclusion Criteria:

* Complete spinal lesion or complete bilateral lesion of sacral / pudendal nerves.
* Degenerative disease of the central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spinelli, MD, Principal Investigator — Ospedale Niguarda Ca' Granda, Milan, Italy; Karel Everaert, MD, Principal Investigator — University Ghent; Philip Van Kerrebroeck, MD, Principal Investigator — Academisch Ziekenhuis, Maastricht, The Netherlands; Emmanuel Chartier-Kastler, MD, Principal Investigator — Hôpital de la Pitié Salpétrière, Paris, France; Arndt Van Ophoven, MD, Principal Investigator — Marienhospital Herne Klinikum der Ruhr-Universität, Herne, Germany; Karl Sievert, MD, Principal Investigator — Klinik für Urologie Oberarzt-Sekretariat, Tübingen, Germany; Suzy Elneil, MD, Principal Investigator — National Hospital for Neurology and Neurosurgery, London, UK
Locations (8):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- France (2):
  - Centre Hospitalier Universitaire de Lyon-Sud, Lyon
  - Hôpital de la Pitié Salpétrière, Paris
- Germany (2):
  - Marienhospital Herne, Klinikum der Ruhr-Universitaet Bochum, Herne
  - Klinik für Urologie Oberarzt-Sekretaria, Tübingen
- Niguarda Ospedale Ca' Granda, Milan, Italy
- Academisch Ziekenhuis, Maastricht, Netherlands
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 patients were included in the study: 9 patients did not pass the test stimulation period, 1 patient dropped out due to exclusion criteria, 1 patient dropped out due to protocol deviation during screening visit, 1 patient dropped out before test stimulation due to early termination of the study, leaving 5 patients who were randomized.
Period: Overall Study
Arm/Group | ON / OFF | OFF / ON
Started | 3 | 2
Completed | 1 | 2
Not Completed | 2 | 0
Not completed — early termination of the study | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was based on all randomized patients in the study. Due to early termination of the study, only 17 patients have been enrolled versus 78 planned enrolled patients. No analysis was done comparing the functional bladder capacity between the two intervention groups due to the low patient numbers in each group.
Groups:
- Total Patient: The patient demographic were analysed without splitting by study intervention since all randomized subjects were to receive both stimulation options (ie, ON and OFF)."
Arm/Group | Total Patient
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: year] | 41.60 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  Belgium | 2
  Italy | 1
  United Kingdom | 1
  France | 1

OUTCOME MEASURES:

1. Primary Outcome: Functional Bladder Capacity
Description: Functional Bladder capacity is measured as the average passed volume per episode, in milliliters, as recorded in the patient's voiding diary during the observation period. Due to the small number of patients in each group, the summary on the functional bladder capacity was provided for the combined groups.
Time Frame: Baseline, 4 weeks after implant, 8 weeks after implant
Population: Due the small number of patients in each group, the summary on the functional bladder capacity was provided for the combined groups.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- All Randomized Patients: All randomized patients have been used for the primary objective. Due to the small number of patients in each group, the summary on the functional bladder capacity was provided for the combined groups.
  Combined groups:
  * group ON/OFF :Stimulation ON for 4 weeks, followed by stimulation OFF for 4 weeks
  * group OFF/ON: Stimulation OFF for 4 weeks, followed by stimulation ON for 4 weeks.
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 5
ml
  Baseline | 186.02 (38.15)
  4 weeks after impalnt | 367.16 (201.17)
  8 weeks after implant: number analyzed (Participants) | 3
  8 weeks after implant | 346.07 (177.98)

ADVERSE EVENTS:
Time Frame: Adverse event reporting started at enrollment until study completion and/or study exit, an average of 14 months, whatever applies.
Groups:
- All Enrolled Patients: Adverse events in this study were reported on the 17 enrolled patients. Due to the small number of patients in each group, the summary on adverse events was provided for the combined groups.
Arm/Group | All Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 7/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Patients (N=17)
Infection of the device stimulator (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Patients (N=17)
URINARY INFECTION (Infections and infestations) | 4 (6)
pain after surgery (Surgical and medical procedures) | 1 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Battery empty at 07h30 and return of symptoms (Investigations) | 1 (1)
Lead cut by the nurse (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No